CLINICAL TRIAL: NCT02831647
Title: Tolerance and Acceptability of AYMES PRAGUE
Brief Title: Acceptability and Tolerance Study of New Oral Nutritional Supplement PRAGUE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aymes International Limited (Industry)
Collaborators: Eat Well Now (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AY:AC1
Record Dates: First submitted 2016-07-11; First posted 2016-07-13 (Estimated); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Malnutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- intervention (Experimental): Patients established on an oral nutritional supplement, being prescribed 1-2 oral nutritional supplement (ONS) providing at least 300 kcal/day will be changed onto an equivalent prescription of AYMES PRAGUE for a period of 9 days.
  Interventions: Dietary Supplement: AYMES PRAGUE

INTERVENTIONS:
Dietary Supplement: AYMES PRAGUE — AYMES PRAGUE is a ready to drink, high energy, low volume oral nutritional supplement drink. It provides 300 kcal and 12g protein per 125ml serving. It is a Food for Special Medical Purposes (FSMP) and must therefore be used under medical supervision. It is not designed as a sole source of nutrition.

SUMMARY:
Tolerance and Acceptability of new oral nutritional supplement - AYMES PRAGUE

DETAILED DESCRIPTION:
To evaluate tolerance and acceptability of AYMES PRAGUE in patients requiring supplementary oral nutritional support compared with currently available alternatives, measuring outcomes of GI effects, Compliance, product preference,convenience etc.

To obtain data to support an ACBS submissions for AYMES PRAGUE (to allow for prescription in the community at NHS expense).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years) who are able to communicate their views regarding acceptability.
* Patients established on an oral nutritional supplement, being prescribed 1-2 ONS providing approximately 300kcal/day
* Patients expected to require oral nutritional supplementation for at least 2 further weeks.
* Informed consent obtained.

Exclusion Criteria:

* Participation in any other studies involving investigational or marketed products concomitantly or within two weeks prior to entry into the study
* Patients requiring a milk-free diet
* Patients with medical or dietary contraindication to any feed ingredients (see appendix 2 of protocol for full list)
* Patients with significant renal or hepatic impairment
* Patients with swallowing impairment requiring thickened fluids
* Patients with inflammatory bowel disease or previous bowel resection.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
GI side effects when using AYMES PRAGUE | 9 DAYS
  Recording of absence/presence of any nausea, vomiting, abdominal pain, bloating / flatulence, when using AYMES PRAGUE as assessed by presence / absence of side effect compared to baseline period

SECONDARY OUTCOMES:
Change to bodyweight of subjects when using AYMES PRAGUE | 9 days
  Recording of bodyweight (in kg) at start of study, start of intervention and end of intervention for comparison to investigate any trend in weight change during the intervention period compared to baseline
Compliance with prescription of AYMES PRAGUE | 9 days
  Recording of amount of AYMES PRAGUE consumed by subjects compared to amount prescribed. Good compliance = >80% of prescribed being consumed. Same data collected for baseline product and compared with that of AYMES PRAGUE
Bowel habits of subjects when using AYMES PRAGUE - frequency | 9 days
  Recording of bowel habits whilst subjects consuming AYMES PRAGUE, as assessed by frequency of bowel movements (number of stools per day) and compared to same data recorded during baseline period
Bowel habits of subjects when using AYMES PRAGUE - stool consistency | 9 days
  Recording of bowel habits whilst subjects consuming AYMES PRAGUE, as assessed by consistency of stools (assessed by Bristol Stool Chart) and compared to same data recorded during baseline period

IPD SHARING:
Plan to Share IPD: No